CLINICAL TRIAL: NCT04037982
Title: A Randomized Controlled Study on the Safety of Total Laparoscopy and Traditional Open Pancreaticoduodenectomy in the Treatment of Periampullary Tumors
Brief Title: RCT Study on Safety of LPD and OPD in the Treatment of Periampullary Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Chief Physician, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-LPD
Record Dates: First submitted 2019-07-28; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Periampullary Tumor; Complication; Death; Survival
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPD (Experimental): In this group, patients will undergo laparoscopic pancreaticoduodenectomy.
  Interventions: Procedure: laparoscopic pancreaticoduodenectomy
- OPD (Active Comparator): In this group, patients will undergo open pancreaticoduodenectomy.
  Interventions: Procedure: Open pancreaticoduodenectomy

INTERVENTIONS:
Procedure: laparoscopic pancreaticoduodenectomy — During laparoscopic surgery, the surgeon makes several smaller incisions in your abdomen and inserts special instruments, including a camera that transmits video to a monitor in the operating room. The surgeon watches the monitor to guide the surgical tools in performing the Whipple procedure. Laparoscopic surgery is a type of minimally invasive surgery.
  Arms: LPD
Procedure: Open pancreaticoduodenectomy — During an open procedure, your surgeon makes an incision in your abdomen in order to access your pancreas. This is the most common approach and the most studied.
  Arms: OPD

SUMMARY:
Pancreaticoduodenectomy (PD) is considered one of the most complex and dangerous procedures in general surgery. This procedure is the preferred surgical procedure for treating tumors around the ampulla. Traditional open pancreaticoduodenectomy (OPD) has brought great surgical trauma to patients while treating diseases. In 1994, Gagner et al first reported laparoscopic pancreaticoduodenectomy (LPD). With the development of laparoscopic techniques, the updating of devices, and the continuous accumulation of laparoscopic gastrointestinal surgery experience, the results of retrospective studies published show that there is no significant difference in safety between LPD and OPD. However, the results of the recently published RCT study show that the mortality associated with LPD complications is five times greater than that of OPD. At present, the security of LPD has been controversial. Therefore we conducted a prospective randomized controlled trial with a primary outcome of perioperative complications, providing evidence-based results for the safe and effective clinical development of LPD.

ELIGIBILITY:
Preoperative imaging diagnosis of periampullary tumor, or preoperative pathological diagnosis of periampullary tumor, preoperative evaluation can be performed pancreaticoduodenectomy; Serum bilirubin was less than 100 μ mol/L before operation; Sign a written informed consent form and agree to be randomly divided into groups for surgical treatment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | 30 days after operation
  The patients number with complications / The total number in this group

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR